CLINICAL TRIAL: NCT06074536
Title: Impact of Training in the Patient-centered Approach on Shared Decision-making in the Colorectal Cancer Screening: a Cluster Randomized Trial
Brief Title: Impact of Training Patient-centered Approach on Shared Decision in Colorectal Cancer Screening
Acronym: FACELE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CNGE Conseil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CNGE-2021-04; IDRCB:2023-A00859-36 (Other: ANSM)
Record Dates: First submitted 2023-09-21; First posted 2023-10-10 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer Screening

STUDY DESIGN:
Intervention Model Description: Patient-centered face-to-face training for General Practitioners on implementation of a shared decision
Who Masked: Participant
Masking Description: Patient not informed of the randomization arm to which their general practitioner enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): The recruited GPs will be randomized into 2 parallel groups (interventional and control). Following this randomization, the GPs from the interventional group will undergo face-to-face training to the patient-centered approach.
  Interventions: Procedure: patient-centered approach training
- Control arm (No Intervention): The GPs of the control group will take care the patient according to current screening recommendations and procedures organized by the colorectal cancer (CCR) mass screening.

INTERVENTIONS:
Procedure: patient-centered approach training — face to face training of general practitioner of interventional arm
  Arms: Interventional arm

SUMMARY:
The purpose of this study is to compare the effect of face-to-face training of general practitioners on the implementation of a shared decision (in the context of colorectal cancer screening), versus current practice (i.e. without training in the patient-centered approach).

DETAILED DESCRIPTION:
Colorectal cancer (CRC) affects 95% of cases of people aged over 50 years old with an average age of diagnosis of 71 years for men and 73 years for women with a higher prevalence in women. By the age of 75, 4 out of 100 men and 3 out of 100 women will have developed colorectal cancer.

In France, CRC screening is based on a guaiac faecal occult blood test in subjects at risk average, carried out every 2 years from 50 to 74 years old. In the event of a positive test, a colonoscopy should be performed. Participation in the programme colorectal cancer screening has been declining since 2016-2017.

The implementation of screening faces many barriers on the physian's side and/or on the patient's side. During of the last 2020-2021 screening campaign, only 6.1 million people took a screening test, which represented a participation rate of 28.9%, while it is commonly admitted that a screening rate >50% would be necessary to reduce CRC mortality.

Some barriers are specific to CRC screening. for patient, reluctance to carry out screening, analysis of stools, and fear of cancer. For the physian, the discomfort in approaching screening and the uncertainty of the relevance of the test for some patients. The know-how and quality of information and communication with patients is at the forefront.

Physian must adapt their communication to the possibilities understanding of the subject to explain, convince, and bring the patient to carry out screening. Active listening is a technique particularly suitable for adopting a person-centred approach making it possible to take into account the patient perspectives in order to arrive at a shared decision.

This most often involves helping and giving the patient the means to manage their problems, involving them in a prevention project (non-requesting patient) or supporting them and motivating them in their approach (requesting patient).

The hypothesize of this study is that training general practitioners in a patient-centered approach will enable the implementation of greater shared decision-making work with the patient during a CRC screening presentation consultation.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 50 to 74:
* Eligible for organized CRC screening,
* Having declared as attending clinician a general practitioner investigator of the study

  ✓ Consulting their attending clinician for the duration of the study,
* AND able and willing to comply with all trial requirements

Non inclusion Criteria:

- ✓ Screened for CRC less than 2 years ago

* Not eligible for organized CRC screening:

  * History of adenomas or CRC:

    - Family (1st degree)
  * Personal history of IBD:

    * Crohn's disease
    * Ulcerative colitis)
  * Hereditary predispositions:

    * Familial adenomatous polyposis
    * Hereditary non-polyposis colorectal cancer (Lynch syndrome)
* Patient with symptoms requiring colonoscopy
* Having a level of literacy that does not allow the completion of the self-questionnaire.
* Having an inability to give express consent.
* Being under guardianship, curatorship or having cognitive disorders

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-03-06 (Actual); Primary Completion 2027-05-06 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
The Measurement of the achievement oh the shared decision shared decision making in CRC screening using the patient shared a self-decision-making questionnaire (SDM-Q9), validated in French | 6 to 8 months after after patient nclusion (carrying out the screening test)
  comparison of the mean of the SDM-Q9 between each arm of the study from 0 (weak shared decision) to 100 (strong shared decision). We will compare the average of the SDM-Q9 between each arm of the study

SECONDARY OUTCOMES:
Evaluate the effect of training on the CRC screening rate | Measurements taken 6 months after the last patient was included in the trial, i.e. no later than 18 months after the start of the trial
  participation rate in organized CRC screening at individual level. Measurements taken 6 months after the last patient was included in the trial,
Confronting the shared decision made by the patient regarding the completion of CRC screening | Measurements taken 6 months after the last patient was included in the trial, i.e. no later than 18 months after the start of the trial
  Participation rate (IC95%) in CRC screening according to the patient's decision at the end of the initial consultation: wish to be screened, neutral, wish not to be screened.
Explore understanding of the shared decision process among general practitioners and patients | Data collected immediately after the inclusion visit
  Proportion (IC95%) of included patients with a SURE test result of less than 4

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle AUGER-AUBIN, Pr, Study Chair — cabinet de groupe pluriprofessionnel 40 rue Carnot 95230 Soisy-Sous-Montmorency
Locations (1):
- Cabinet de groupe pluriprofessionnel, Soisy-sous-Montmorency, France